CLINICAL TRIAL: NCT06346548
Title: Monocentric Observational Cross-sectional Study on the Chromatic Perception of Digital Systems in Aesthetic Field
Brief Title: Study on the Chromatic Perception of Digital Systems in Aesthetic Field
Status: Completed | Type: Observational
Sponsor: Paolone Gaetano (Other)
Responsible Party: Sponsor-Investigator, Paolone Gaetano, Principal Investigator, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: VF-ES-DIG
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Color Detection of Upper Central Incisors
MeSH Terms: interventions — Photography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: This group will include patients with an age between 18 years old and 29 years old. The recruitment doesn't include a gender selection
  Interventions: Other: oral photography
- Group 2: This group will include patients with an age between 30 years old and 59 years old. The recruitment doesn't include a gender selection
  Interventions: Other: oral photography
- Group 3: This group will include patients with an age over 60 years old. The recruitment doesn't include a gender selection
  Interventions: Other: oral photography

INTERVENTIONS:
Other: oral photography — The patient will under go three different color detecting methods. Two photography methodologies and one intra oral digital scanner
  Other Names: digital intra oral scanner

SUMMARY:
The study under consideration aims to evaluate differences in chromatic perception among three distinct color acquisition methodologies. Specifically, recruited patients will undergo testing with three different color detection systems, including two intraoral photography methodologies and one digital intra oral scanning. All procedures conducted are part of normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good oral health
* Age over 18 years old
* Signing of an informed consent form according to the protocol

Exclusion Criteria:

* Any type of restoration on the upper central and lateral incisors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As part of normal clinical practice, the expected population for the examination (anticipated number of patients = 78) will undergo three different chromatic detection methodologies to assess differences in chromatic perception through intra and inter group analyses. The selected sample will be divided equally only based on three different age groups (18-29 years, 30-59 years, >60 years).
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Comparison of chromatic values of the upper central incisors | 9 months
  Comparison of chromatic values of the upper central incisors (within and between age groups) extracted from the 3 chromatic detection methodologies(intra oral photography, extra oral photography, intra oral digital scanner), aiming to determine any statistical differences.

CONTACTS AND LOCATIONS:
Overall Officials: Paolone Gaetano, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No